CLINICAL TRIAL: NCT03073161
Title: Flavonoid Intake and Periodontal Outcomes After Sanative Therapy
Brief Title: Flavonoid Intake and Periodontal Healing
Status: Completed | Type: Observational
Sponsor: Brock University (Other)
Collaborators: Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery (Other)
Responsible Party: Principal Investigator, Wendy E. Ward, Ph.D., Professor and Canada Research Chair, Brock University
Other Study IDs: 16-114
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Periodontal Attachment Loss; Periodontal Pocket
Keywords: flavonoids; tea; dietary intake; nutritional supplements; periodontal disease; healing; sanative therapy
MeSH Terms: conditions — Periodontal Attachment Loss; Periodontal Pocket; Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva is being collected for before and after sanative therapy for analysis of inflammatory markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Periodontitis is a chronic inflammatory disease that, if untreated, will lead to tooth loss. To treat periodontal disease, sanative therapy is used as a first line cost-effective strategy to manage periodontal disease and thus prevent tooth loss. Diet is emerging as a modifiable factor that may help an individual to more fully respond to treatments such as sanative therapy. Dietary flavonoids, abundant in fruits and tea, may be particularly beneficial. Patients with moderate to severe chronic generalized periodontitis and undergoing sanative therapy will be recruited for the study. Mean clinical attachment loss as well as other clinical measures will be assessed at baseline and 8 to 12 weeks following sanative therapy to measure periodontal healing. At baseline and follow-up appointment, the following will be assessed to examine associations with clinical measures of periodontal healing: intakes of macronutrients and micronutrients, fruits, vegetables and tea as well as supplement use and salivary markers of inflammation.

DETAILED DESCRIPTION:
Periodontitis is a chronic oral infection that results in the breakdown of connective tissue and alveolar bone that support the teeth. Bacteria and the body's own immune system mediate the severity of periodontitis, where teeth may become loose, fall out or have to be removed. Sanative therapy is a non-surgical process invovling mechanical debridement of bacterial biofilms on roots of teeth, below the gum line. A previous study found that a diet higher in fruits and vegetables, beta-carotene, vitamin C, alpha-tocopherol, and fish oils (specifically eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)) was positively associated with periodontal healing after sanative therapy. There is some evidence that higher intakes of flavonoids and thus flavonoid-containing foods may benefit periodontal health. These foods include a wide variety of fruits and tea. The relationship of flavonoid intake within the overall dietary pattern has not been assessed in relation to recovery from sanative therapy and associated markers of improved periodontal health. The overall objective is to determine if higher dietary flavonoid intakes are associated with improved clinical outcomes after sanative therapy compared to individuals with lower intakes. At baseline and the follow-up appointment, the following will be assessed: dietary intakes of macronutrients and micronutrients using the Block 2015 food frequency questionnaire; intakes of fruit, vegetables and fiber using the Block Dietary Fruit-Vegetable-Fiber Screener; nutritional supplement use and tea intake using in specially developed questionnaires and salivary markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing sanative therapy for moderate to severe chronic generalized periodontitis. Chronic periodontitis is classified as generalized if >30% of sites are involved. Severity of periodontitis is based on the amount of clinical attachment loss (CAL) with moderate and severe chronic generalized periodontitis defined as 3 to 4 mm CAL or > 5 mm CAL, respectively.

Exclusion Criteria:

* under 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing sanative therapy for the treatment of moderate to severe chronic generalized periodontitis.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Loss (CAL) (also called Periodontal Attachment Loss) | At baseline and at follow-up (8 to 12 weeks after completion of sanative therapy)
  Periodontal healing is evaluated based on changes in clinical attachment loss (mm)

SECONDARY OUTCOMES:
Probing Depth | At baseline and at follow-up (8 to 12 weeks after completion of sanative therapy)
  Periodontal healing is evaluated based on changes in probing depth (mm)
Bleeding on Probing | At baseline and at follow-up (8 to 12 weeks after completion of sanative therapy)
  Inflammation is determined by percent of bleeding sites that are measured at 6 sites per tooth
Plaque Index | At baseline and at follow-up (8 to 12 weeks after completion of sanative therapy)
  O'Leary Plaque Score Index is a score of the total amount of plaque present at 4 surfaces of a tooth

OTHER OUTCOMES:
Dietary Nutrient Intakes | Completed at baseline and follow-up (8 to 12 weeks after completion of sanative therapy)
  Dietary intakes measured using the BLOCK food frequency questionnaire
Tea Intakes | Completed at baseline and follow-up (8 to 12 weeks after completion of sanative therapy)
  Quantity of tea and type of tea consumed will be determined using a questionnaire
Servings of fruits, vegetables and fibre | Completed at baseline and follow-up (8 to 12 weeks after completion of sanative therapy)
  A questionnaire called the Block Fruit-Vegetable-Fiber Screener is used to provide a score that pertains to number of servings of fruits, vegetables and fiber consumed over past month
Dietary Supplement Intakes | Completed at baseline and follow-up (8 to 12 weeks after completion of sanative therapy)
  Intakes of specific dietary supplements measured using a dietary supplement questionnaire
Salivary Markers of Inflammation | Measured at baseline and follow-up (8 to 12 weeks after completion of sanative therapy)
  Specific markers of inflammation measured in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Wendy E Ward, Ph.D., Principal Investigator — Brock University
Locations (1):
- Dr. Peter C. Fritz, Reconstructive Periodontics and Implant Surgery, Fonthill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No